CLINICAL TRIAL: NCT06840041
Title: The Relationship Between Vaginal Microbiota and Post-Cesarean Section Wound Infection
Brief Title: Vaginal Microbiota and Post-cesarean SSI
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Other Study IDs: Obst19225
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Site Infection; Cesarean Section; Complications, Wound, Infection (Following Delivery)
Keywords: cesarean section; SSI; vaginal microbiota
MeSH Terms: conditions — Wounds and Injuries; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cesarean section group: This observational study will enroll 160 women undergoing cesarean section. Participants will provide vaginal swab samples for culture, both pre-operatively and post-operatively. They will be monitored post-operatively for the development of wound infections, with wound assessments performed according to standard clinical practice. Demographic and clinical data, including antibiotic use, gestational age, and comorbidities, will be collected to assess the relationship between vaginal microbiota and post-cesarean wound infections.
  Interventions: Diagnostic Test: Vaginal swab and culture

INTERVENTIONS:
Diagnostic Test: Vaginal swab and culture — Participants will undergo vaginal swab collection both pre-operatively, immediately prior to the cesarean section, and post-operatively, within a defined timeframe after the procedure. The swabs will be collected using sterile swabs, following standardized procedures to ensure accurate sampling of the vaginal microbiota. The collected samples will then be sent to a designated laboratory for culture and analysis. This process will identify and characterize the bacterial composition of the vaginal microbiota, allowing researchers to investigate potential correlations between specific microbial profiles and the development of post-cesarean section wound infections

SUMMARY:
The goal of this observational study is to investigate the relationship between vaginal microbiota composition and the development of post-cesarean section wound infection in women undergoing cesarean delivery. The main question it aims to answer is:

Is there a correlation between specific vaginal microbiota profiles and the incidence of post-cesarean section wound infection? Can specific bacterial taxa or diversity indices within the vaginal microbiota predict the risk of post-cesarean section wound infection?

Participants will:

Provide vaginal swab samples pre-operatively and post-operatively. Undergo standard post-cesarean section care and follow-up. Have wound assessment performed per standard of care, and have data collected regarding wound infection status.

Have demographic and clinical data collected, including but not limited to, antibiotic use, gestational age, and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing elective or emergency cesarean section (CS).
* Singleton pregnancy.
* Cesarean section performed at ≥ 37 weeks of gestation.

Exclusion Criteria:

* Use of antibiotics within two weeks prior to delivery.
* Known immunodeficiency.
* Chronic infections.
* Ruptured membranes for more than 18 hours.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is exclusively for female participants undergoing cesarean section. Biological females are the only eligible participants due to the focus on vaginal microbiota and its relationship to post-cesarean section wound infections.
Study Population: This study will enroll pregnant women undergoing either elective or emergency cesarean section at or beyond 37 weeks of gestation. Participants must have a singleton pregnancy. Women with known immunodeficiency, chronic infections, or those who have received antibiotics within two weeks prior to delivery will be excluded. Additionally, women with ruptured membranes for more than 18 hours will be excluded to minimize the potential influence of prolonged exposure to mixed flora. The study aims to investigate the relationship between vaginal microbiota and post-cesarean section wound infection within this defined population.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of Vaginal Microbiota Composition and Surgical Site Infection (SSI) Incidence | 4 weeks after the surgery.
  This outcome will assess the differences in vaginal microbiota composition between women who develop a surgical site infection (SSI) following cesarean section and those who do not. Microbiota composition will be determined through culture and analysis of vaginal swab samples collected pre-operatively and post-operatively. Comparisons will focus on identifying significant variations in bacterial taxa, diversity indices, and overall microbial community structure between the two groups.

SECONDARY OUTCOMES:
Predictive Value of Specific Vaginal Bacterial Species for Surgical Site Infection (SSI). | 6 months
  This outcome will evaluate the ability of specific bacterial species identified in vaginal swab samples to predict the development of surgical site infection (SSI) following cesarean section. Logistic regression analysis will be used to determine the independent predictive value of individual bacterial species, as well as combinations of species, for SSI. The analysis will assess the odds ratios, confidence intervals, and p-values associated with each bacterial species.

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed Alhagrasy, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified Individual Participant Data (IPD) that underlie the results reported in this article, including study protocol, statistical analysis plan, and analytic code, will be made available upon reasonable request to qualified researchers after publication. Requests should be submitted to MuhamedAhmed.216@azhar.edu.eg. Proposals will be reviewed by the Department of Obstetrics and Gynecology, Al-Azhar University to ensure that the proposed use of the data is scientifically sound and ethical. Data will be shared in a secure, password-protected format, and a data sharing agreement will be required to ensure responsible use and protection of participant confidentiality. The data will be available for 5 years following publication. Publication of results will be made without identifiers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years after publication.
Access Criteria: Access to de-identified Individual Participant Data (IPD) will be granted to qualified researchers with a demonstrated scientific need and a clearly defined research question. Researchers must submit a formal request to MuhamedAhmed.216@azhar.edu.eg, outlining their research proposal, including the specific data requested, the intended use of the data, and their qualifications. Requests will be reviewed by the Department of Obstetrics and Gynecology, Al-Azhar University to ensure scientific merit and ethical compliance. Researchers must agree to sign a data sharing agreement that outlines the terms of data use, including restrictions on redistribution and requirements for appropriate data security and confidentiality.